CLINICAL TRIAL: NCT06991712
Title: Comparisons of Nicotinamide Adenine Dinucleotide (NAD) Precursors for Neuroenhancement in Glaucoma Patients
Brief Title: Comparisons of NAD Precursors for Neuroenhancement in Glaucoma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christopher Kai Shun Leung (Other)
Responsible Party: Sponsor-Investigator, Christopher Kai Shun Leung, Chairperson and Clinical Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H029
Record Dates: First submitted 2025-05-16; First posted 2025-05-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Glaucoma
Keywords: NAD Precursor; Nicotinic Acid; Nicotinamide; Nicotinamide Mononucleotide; Nicotinamide Riboside
MeSH Terms: conditions — Glaucoma | interventions — nicotinamide-beta-riboside; Niacinamide; Nicotinamide Mononucleotide; Niacin; Starch

STUDY DESIGN:
Intervention Model Description: NR, NAM, NMN, or NA in mole equivalent amount, or placebo, will be randomly assigned to 138 patients, 23 per group (a total of 4 treatment groups and 2 placebo groups). Each patient will receive a daily dose of 300 mg NR, 125 mg NAM, 350 mg NMN, 125 mg NA or 300 mg placebo (corn starch capsule) at 9 am each day for two weeks. The study will be conducted in 2 phases. In Phase I, participants will be randomized to placebo, NR, or NAM. In Phase II, participants will be randomized to receive, placebo, NA, or NMN.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, investigators, the outcome assessors, and data analysts will be masked before and after assignment to intervention.
  The subject will be unmasked as per of the request of Principal Investigator in case of serious adverse event or if emergency unblinding is deemed essential for clinical management. All instances of the unblinding will be documented in the study binder. Unmasked subject will exit from the study and resumes normal clinical management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Nicotinamide Riboside (Phase I) (Experimental)
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Nicotinamide (Phase I) (Active Comparator)
  Interventions: Dietary Supplement: Nicotinamide
- Nicotinamide Mononucleotide (Phase II) (Active Comparator)
  Interventions: Dietary Supplement: Nicotinamide Mononucleotide
- Nicotinic Acid (Phase II) (Active Comparator)
  Interventions: Dietary Supplement: Nicotinic Acid
- Placebo (Phase I) (Placebo Comparator)
  Interventions: Other: Placebo (Corn Starch)
- Placebo (Phase II) (Placebo Comparator)
  Interventions: Other: Placebo (Corn Starch)

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Oral supplementation of 300mg Nicotinamide Riboside (NR) daily for 2 weeks
  Other Names: NR
  Arms: Nicotinamide Riboside (Phase I)
Dietary Supplement: Nicotinamide — Oral supplementation of 125mg Nicotinamide/Niacinamide (NAM) daily for 2 weeks
  Other Names: Niacinamide; NAM
  Arms: Nicotinamide (Phase I)
Dietary Supplement: Nicotinamide Mononucleotide — Oral supplementation of 350mg Nicotinamide Mononucleotide (NMN) daily for 2 weeks
  Other Names: NMN
  Arms: Nicotinamide Mononucleotide (Phase II)
Dietary Supplement: Nicotinic Acid — Oral supplementation of 350mg Nicotinic Acid (NA) daily for 2 weeks
  Arms: Nicotinic Acid (Phase II)
Other: Placebo (Corn Starch) — Oral supplementation of 300mg Placebo daily for 2 weeks
  Arms: Placebo (Phase I)
Other: Placebo (Corn Starch) — Oral supplementation of 300mg Placebo daily for 2 weeks
  Arms: Placebo (Phase II)

SUMMARY:
The goal of this clinical trial is to determine whether oral supplementation with different nicotinamide adenine dinucleotide (NAD) precursors can improve visual function in adults with primary open-angle glaucoma. The main questions it aims to answer are:

1. Does daily oral administration of equimolar doses of nicotinamide riboside (NR), nicotinamide (NAM), nicotinamide mononucleotide (NMN), or nicotinic acid (NA) improve visual field sensitivity in glaucoma patients over the short term?
2. How do plasma NAD+ metabolite profiles change after administration of each precursor, and do these changes relate to improvements in visual function?

Researchers will compare NR, NAM, NMN, NA, and placebo groups to see if any of the NAD precursors lead to greater improvements in visual field sensitivity or changes in blood NAD+ metabolite levels compared to placebo.

Participants will:

Be randomly assigned to receive one of the four NAD precursors or placebo daily for two weeks.

Undergo comprehensive eye examinations, including visual field testing and optical coherence tomography, at baseline and after two weeks.

Provide blood samples before and after the intervention for measurement of NAD+ metabolites.

Have safety monitored through clinical examination.

This study will help identify whether boosting NAD+ levels with specific precursors offers functional benefit in glaucoma, and which blood metabolites may mediate these effects.

DETAILED DESCRIPTION:
This prospective randomized, double-blind, placebo-controlled clinical trial evaluates four nicotinamide adenine dinucleotide (NAD) precursors for neuroenhancement in 138 adults with primary open-angle glaucoma. Participants are randomly assigned to receive daily oral supplementation for one week with equimolar doses of nicotinamide riboside (300 mg), nicotinamide (125 mg), nicotinamide mononucleotide (350 mg), nicotinic acid (125 mg), or placebo. The study assesses short-term changes in visual field sensitivity using Humphrey Field Analyzer 24-2 testing and measures NAD+ metabolite profiles through liquid chromatography-tandem mass spectrometry (LC-MS/MS) and gas chromatography-tandem mass spectrometry (GC-MS/MS) analysis of plasma and peripheral blood mononuclear cells collected at baseline, pre-dose, and post-dose timepoints.

Secondary objectives include comparing pattern electroretinogram nerve fiber layer thickness measurements before and after treatment and analyzing correlations between systemic NAD+ metabolite elevations and functional visual improvements. Blood samples undergo standardized processing with Lymphoprep separation, snap-freezing, and derivatization protocols prior to mass spectrometry analysis using Agilent and Thermo Fisher systems with predefined NAD+ metabolite inclusion lists.

Statistical analysis employs linear mixed models to compare within-group and between-group changes, with intention-to-treat principles. The study design addresses gaps in comparative NAD precursor bioavailability data by testing equimolar doses in a targeted glaucoma population, while maintaining double-blinding through computer-generated randomization and masked outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma patients
* age ≥ 18 years
* best corrected VA ≥20/40
* IOP <21 mmHg
* visual field mean deviation better than -24 dB on standard automated perimetry 24-2 SITA standard

Exclusion Criteria:

* pathological myopia
* diseases that may cause visual field loss or optic disc abnormalities other than glaucoma
* inability to perform reliable visual field
* suboptimal quality of OCT images
* diabetic retinopathy/maculopathy
* history of abnormal liver function within 12 months
* known allergy to NAD precursor supplement(s)
* pregnancy or lactation
* use of NAD precursor supplements 14 days prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in visual field sensitivity | 2 weeks
  Visual field will be measured with automated static perimetry by the Humphrey Field Analyzer 3 24-2 SITA standard strategy (HFA; Carl Zeiss Meditec). Two reliable visual fields will be obtained for each eye at the baseline examination, with at least 10 minutes of rest in between, and two reliable visual fields will be obtained for each eye at week two.
  Change in visual field index (VFI) and threshold sensitivity (dB) before and two weeks after intervention between treatment groups will be compared.

SECONDARY OUTCOMES:
Blood NA and NAD+ metabolome | 2 weeks
  At baseline, plasma and PBMC samples will be collected on the day of VF test before the intake of NAD precursor or placebo between 9am and 10am. After two weeks of oral administration of NAD+ precursor or placebo, two blood samples will be collected: between 9 am and 10 am (pre-dose), and then between 11am and 12 noon (post-dose). The sample will be processed by liquid chromatography-tandem mass spectrometry (LC-MS/MS) and chromatography-tandem mass spectrometry (GC-MS/MS) to measure the amounts of NAD+ metabolites. Changes in NAD metabolites before and 2 weeks after intake of NAD precursors will be compared between treatment groups.
Change in pattern ERG measurements | 2 weeks
  Pattern Electroretinogram (PERG) will also be performed at baseline and follow-up for every other subject included in the study. Changes in PERG measurements including P50 and N95 amplitudes, before and two weeks after intervention, will be compared between the placebo group and the NAD precursor group.
Retinal nerve fiber layer thickness and defect imaging by optical coherence tomography | 2 weeks
  At baseline and week two follow-up visits, RNFL imaging will be performed with the Cirrus HD-OCT (Carl Zeiss Meditec) using the optic nerve head (6x6 mm2) cube scan covering both the macula and the parapapillary area (512x256 pixels). Changes in average RNFL thickness before and two weeks after intervention will be compared between treatment groups.

OTHER OUTCOMES:
Impact of age on the change in visual field sensitivity | 2 weeks
  To investigate whether age is associated with change in VF sensitivities

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kai-shun LEUNG, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- HKU Eye Centre, Wong Chuk Hang, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allison K, Patel D, Alabi O. Epidemiology of Glaucoma: The Past, Present, and Predictions for the Future. Cureus. 2020 Nov 24;12(11):e11686. doi: 10.7759/cureus.11686. PMID 33391921
- [Background] Bengtsson B, Lindgren A, Heijl A, Lindgren G, Asman P, Patella M. Perimetric probability maps to separate change caused by glaucoma from that caused by cataract. Acta Ophthalmol Scand. 1997 Apr;75(2):184-8. doi: 10.1111/j.1600-0420.1997.tb00121.x. PMID 9197570
- [Background] Bledi Petriti, Alessandro Rabiolo, Pete Williams, Kai-Yin Chau, Gerassimos Lascaratos, David F Garway-Heath; Primary open angle glaucoma patients have lower systemic mitochondrial function, associated with lower systemic nicotinamide adenine dinucleotide (NAD) levels, compared to Controls. Invest. Ophthalmol. Vis. Sci. 2023;64(8):483.
- [Background] Bledi Petriti, Gerassimos Lascaratos, David Chau, Williams Peter, David F Garway-Heath; Preliminary data show Normal Tension Glaucoma patients have lower systemic nicotinamide adenine dinucleotide (NAD+) levels and mitochondrial function compared to Controls. Invest. Ophthalmol. Vis. Sci. 2021;62(8):1765.
- [Background] Capuzzi DM, Guyton JR, Morgan JM, Goldberg AC, Kreisberg RA, Brusco OA, Brody J. Efficacy and safety of an extended-release niacin (Niaspan): a long-term study. Am J Cardiol. 1998 Dec 17;82(12A):74U-81U; discussion 85U-86U. doi: 10.1016/s0002-9149(98)00731-0. PMID 9915666
- [Background] Christopher Kai-Shun Leung, Philip Guo, Marco Yu, Gilda Lai; Nicotinamide Riboside for Progressing Glaucoma: A Double-blind, Parallel Group, Randomized, Placebo-controlled Trial - A Report on Neuroenhancement. Invest. Ophthalmol. Vis. Sci. 2023;64(8):4349.
- [Background] Cros C, Cannelle H, Laganier L, Grozio A, Canault M. Safety evaluation after acute and sub-chronic oral administration of high purity nicotinamide mononucleotide (NMN-C(R)) in Sprague-Dawley rats. Food Chem Toxicol. 2021 Apr;150:112060. doi: 10.1016/j.fct.2021.112060. Epub 2021 Feb 12. PMID 33587977
- [Background] De Moraes CG, John SWM, Williams PA, Blumberg DM, Cioffi GA, Liebmann JM. Nicotinamide and Pyruvate for Neuroenhancement in Open-Angle Glaucoma: A Phase 2 Randomized Clinical Trial. JAMA Ophthalmol. 2022 Jan 1;140(1):11-18. doi: 10.1001/jamaophthalmol.2021.4576. PMID 34792559
- [Background] European Food Safety Authority. Tolerable Upper Intake Levels for Vitamins and Minerals (2006). Parma, Italy: European Food Safety Authority; 2006.
- [Background] Medeiros FA, Zangwill LM, Bowd C, Mansouri K, Weinreb RN. The structure and function relationship in glaucoma: implications for detection of progression and measurement of rates of change. Invest Ophthalmol Vis Sci. 2012 Oct 5;53(11):6939-46. doi: 10.1167/iovs.12-10345. PMID 22893677
- [Background] Gardiner SK, Crabb DP. Frequency of testing for detecting visual field progression. Br J Ophthalmol. 2002 May;86(5):560-4. doi: 10.1136/bjo.86.5.560. PMID 11973255
- [Background] Garway-Heath DF, Crabb DP, Bunce C, Lascaratos G, Amalfitano F, Anand N, Azuara-Blanco A, Bourne RR, Broadway DC, Cunliffe IA, Diamond JP, Fraser SG, Ho TA, Martin KR, McNaught AI, Negi A, Patel K, Russell RA, Shah A, Spry PG, Suzuki K, White ET, Wormald RP, Xing W, Zeyen TG. Latanoprost for open-angle glaucoma (UKGTS): a randomised, multicentre, placebo-controlled trial. Lancet. 2015 Apr 4;385(9975):1295-304. doi: 10.1016/S0140-6736(14)62111-5. Epub 2014 Dec 19. PMID 25533656
- [Background] GRAS No 635, available at https://www.accessdata.fda.gov/scripts/fdcc/index.cfm?set=GRASNotices&id=635
- [Background] Gupta D, Chen PP. Glaucoma. Am Fam Physician. 2016 Apr 15;93(8):668-74. PMID 27175839
- [Background] Harwerth RS, Carter-Dawson L, Shen F, Smith EL 3rd, Crawford ML. Ganglion cell losses underlying visual field defects from experimental glaucoma. Invest Ophthalmol Vis Sci. 1999 Sep;40(10):2242-50. PMID 10476789
- [Background] Heijl A, Bengtsson B, Hyman L, Leske MC; Early Manifest Glaucoma Trial Group. Natural history of open-angle glaucoma. Ophthalmology. 2009 Dec;116(12):2271-6. doi: 10.1016/j.ophtha.2009.06.042. Epub 2009 Oct 24. PMID 19854514
- [Background] Hui F, Tang J, Williams PA, McGuinness MB, Hadoux X, Casson RJ, Coote M, Trounce IA, Martin KR, van Wijngaarden P, Crowston JG. Improvement in inner retinal function in glaucoma with nicotinamide (vitamin B3) supplementation: A crossover randomized clinical trial. Clin Exp Ophthalmol. 2020 Sep;48(7):903-914. doi: 10.1111/ceo.13818. Epub 2020 Jul 28. PMID 32721104
- [Background] Institute of Medicine (IOM, 1998). Niacin: In: Dietary Reference Intakes for Thiamin, Riboflavin, Niacin, Vitamin B(6), Folate, Vitamin B(12), Pantothenic Acid, Biotin, and Choline. (National Academy of Sciences/NAS, Institute of Medicine/IOM, Food and Nutrition Board/FNB, Standing Committee on the Scientific Evaluation of Dietary Reference Intakes and its Panel on Folate, Other B Vitamins, and Choline, and the Subcommittee on Upper Reference Levels of Nutrients). Washington (DC): National Academy Press (NAP), pp. 123-149. Available at:http://www.nap.edu/openbook.php?record_id=6015&page=123
- [Background] Ito, T. K., Sato, T., Hakamata, A., Onoda, Y., Sato, S., Yamazaki, F., Horikawa, M., Takahashi, Y., Kitamoto, T., Suzuki, M., Uchida, S., Odagiri, K., & Setou, M. (2020). A nonrandomized study of single oral supplementation within the daily tolerable upper level of nicotinamide affects blood nicotinamide and NAD+ levels in healthy subjects. Translational Medicine of Aging, 4, 45-54. https://doi.org/10.1016/j.tma.2020.04.002
- [Background] Ito, Takashi & Sato, Tomohito & Takanashi, Yusuke & Tamannaa, Zinat & Kitamoto, Takuya & Odagiri, Keiichi & Setou, Mitsutoshi. (2021). A single oral supplementation of nicotinamide within the daily tolerable upper level increases blood NAD+ levels in healthy subjects. Translational Medicine of Aging. 5. 10.1016/j.tma.2021.09.001.
- [Background] Jadeja RN, Thounaojam MC, Bartoli M, Martin PM. Implications of NAD+ Metabolism in the Aging Retina and Retinal Degeneration. Oxid Med Cell Longev. 2020 May 9;2020:2692794. doi: 10.1155/2020/2692794. eCollection 2020. PMID 32454935
- [Background] Kamanna VS, Ganji SH, Kashyap ML. The mechanism and mitigation of niacin-induced flushing. Int J Clin Pract. 2009 Sep;63(9):1369-77. doi: 10.1111/j.1742-1241.2009.02099.x. PMID 19691622
- [Background] Lautrup S, Sinclair DA, Mattson MP, Fang EF. NAD+ in Brain Aging and Neurodegenerative Disorders. Cell Metab. 2019 Oct 1;30(4):630-655. doi: 10.1016/j.cmet.2019.09.001. PMID 31577933
- [Background] Leung CKS, Ye C, Weinreb RN, Yu M, Lai G, Lam DS. Impact of age-related change of retinal nerve fiber layer and macular thicknesses on evaluation of glaucoma progression. Ophthalmology. 2013 Dec;120(12):2485-2492. doi: 10.1016/j.ophtha.2013.07.021. Epub 2013 Aug 30. PMID 23993360
- [Background] Lin C, Mak H, Yu M, Leung CK. Trend-Based Progression Analysis for Examination of the Topography of Rates of Retinal Nerve Fiber Layer Thinning in Glaucoma. JAMA Ophthalmol. 2017 Mar 1;135(3):189-195. doi: 10.1001/jamaophthalmol.2016.5111. PMID 28152147
- [Background] Lin JB, Kubota S, Ban N, Yoshida M, Santeford A, Sene A, Nakamura R, Zapata N, Kubota M, Tsubota K, Yoshino J, Imai SI, Apte RS. NAMPT-Mediated NAD(+) Biosynthesis Is Essential for Vision In Mice. Cell Rep. 2016 Sep 27;17(1):69-85. doi: 10.1016/j.celrep.2016.08.073. PMID 27681422
- [Background] Mahmoudinezhad G, Moghimi S, Proudfoot JA, Brye N, Nishida T, Yarmohammadi A, Kamalipour A, Zangwill LM, Weinreb RN. Effect of Testing Frequency on the Time to Detect Glaucoma Progression With Optical Coherence Tomography (OCT) and OCT Angiography. Am J Ophthalmol. 2023 Jan;245:184-192. doi: 10.1016/j.ajo.2022.08.030. Epub 2022 Sep 10. PMID 36096181
- [Background] Mehmel M, Jovanovic N, Spitz U. Nicotinamide Riboside-The Current State of Research and Therapeutic Uses. Nutrients. 2020 May 31;12(6):1616. doi: 10.3390/nu12061616. PMID 32486488
- [Background] Meyers CD, Carr MC, Park S, Brunzell JD. Varying cost and free nicotinic acid content in over-the-counter niacin preparations for dyslipidemia. Ann Intern Med. 2003 Dec 16;139(12):996-1002. doi: 10.7326/0003-4819-139-12-200312160-00009. PMID 14678919
- [Background] Morgan JM, Capuzzi DM, Guyton JR. A new extended-release niacin (Niaspan): efficacy, tolerability, and safety in hypercholesterolemic patients. Am J Cardiol. 1998 Dec 17;82(12A):29U-34U; discussion 39U-41U. doi: 10.1016/s0002-9149(98)00732-2. PMID 9915660
- [Background] Nouri-Mahdavi K, Nassiri N, Giangiacomo A, Caprioli J. Detection of visual field progression in glaucoma with standard achromatic perimetry: a review and practical implications. Graefes Arch Clin Exp Ophthalmol. 2011 Nov;249(11):1593-616. doi: 10.1007/s00417-011-1787-5. Epub 2011 Aug 26. PMID 21870086
- [Background] Norquist JM, Watson DJ, Yu Q, Paolini JF, McQuarrie K, Santanello NC. Validation of a questionnaire to assess niacin-induced cutaneous flushing. Curr Med Res Opin. 2007 Jul;23(7):1549-60. doi: 10.1185/030079907x199637. PMID 17559750
- [Background] Nouri-Mahdavi K, Hoffman D, Gaasterland D, Caprioli J. Prediction of visual field progression in glaucoma. Invest Ophthalmol Vis Sci. 2004 Dec;45(12):4346-51. doi: 10.1167/iovs.04-0204. PMID 15557442
- [Background] Okabe K, Yaku K, Uchida Y, Fukamizu Y, Sato T, Sakurai T, Tobe K, Nakagawa T. Oral Administration of Nicotinamide Mononucleotide Is Safe and Efficiently Increases Blood Nicotinamide Adenine Dinucleotide Levels in Healthy Subjects. Front Nutr. 2022 Apr 11;9:868640. doi: 10.3389/fnut.2022.868640. eCollection 2022. PMID 35479740
- [Background] Pardue MT, Allen RS. Neuroprotective strategies for retinal disease. Prog Retin Eye Res. 2018 Jul;65:50-76. doi: 10.1016/j.preteyeres.2018.02.002. Epub 2018 Feb 23. PMID 29481975
- [Background] Paolini JF, Mitchel YB, Reyes R, Thompson-Bell S, Yu Q, Lai E, Watson DJ, Norquist JM, Sisk CM, Bays HE. Measuring flushing symptoms with extended-release niacin using the flushing symptom questionnaire: results from a randomised placebo-controlled clinical trial. Int J Clin Pract. 2008 Jun;62(6):896-904. doi: 10.1111/j.1742-1241.2008.01739.x. Epub 2008 Apr 10. PMID 18410350
- [Background] Petriti B, Williams PA, Lascaratos G, Chau KY, Garway-Heath DF. Neuroprotection in Glaucoma: NAD+/NADH Redox State as a Potential Biomarker and Therapeutic Target. Cells. 2021 Jun 5;10(6):1402. doi: 10.3390/cells10061402. PMID 34198948
- [Background] Pirinen E, Auranen M, Khan NA, Brilhante V, Urho N, Pessia A, Hakkarainen A, Kuula J, Heinonen U, Schmidt MS, Haimilahti K, Piirila P, Lundbom N, Taskinen MR, Brenner C, Velagapudi V, Pietilainen KH, Suomalainen A. Niacin Cures Systemic NAD+ Deficiency and Improves Muscle Performance in Adult-Onset Mitochondrial Myopathy. Cell Metab. 2020 Jun 2;31(6):1078-1090.e5. doi: 10.1016/j.cmet.2020.04.008. Epub 2020 May 7. PMID 32386566
- [Background] Poljsak B, Kovac V, Milisav I. Current Uncertainties and Future Challenges Regarding NAD+ Boosting Strategies. Antioxidants (Basel). 2022 Aug 24;11(9):1637. doi: 10.3390/antiox11091637. PMID 36139711
- [Background] Ramsey KM, Yoshino J, Brace CS, Abrassart D, Kobayashi Y, Marcheva B, Hong HK, Chong JL, Buhr ED, Lee C, Takahashi JS, Imai S, Bass J. Circadian clock feedback cycle through NAMPT-mediated NAD+ biosynthesis. Science. 2009 May 1;324(5927):651-4. doi: 10.1126/science.1171641. Epub 2009 Mar 19. PMID 19299583
- [Background] Rajman L, Chwalek K, Sinclair DA. Therapeutic Potential of NAD-Boosting Molecules: The In Vivo Evidence. Cell Metab. 2018 Mar 6;27(3):529-547. doi: 10.1016/j.cmet.2018.02.011. PMID 29514064
- [Background] Shin JW, Sung KR, Lee J, Kwon J. Factors Associated With Visual Field Progression in Cirrus Optical Coherence Tomography-guided Progression Analysis: A Topographic Approach. J Glaucoma. 2017 Jun;26(6):555-560. doi: 10.1097/IJG.0000000000000680. PMID 28410253
- [Background] Sood A, Arora R. Mechanisms of flushing due to niacin and abolition of these effects. J Clin Hypertens (Greenwich). 2009 Nov;11(11):685-9. doi: 10.1111/j.1559-4572.2008.00050.x. PMID 19878384
- [Background] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815
- [Background] Trammell SA, Schmidt MS, Weidemann BJ, Redpath P, Jaksch F, Dellinger RW, Li Z, Abel ED, Migaud ME, Brenner C. Nicotinamide riboside is uniquely and orally bioavailable in mice and humans. Nat Commun. 2016 Oct 10;7:12948. doi: 10.1038/ncomms12948. PMID 27721479
- [Background] Tribble JR, Otmani A, Sun S, Ellis SA, Cimaglia G, Vohra R, Joe M, Lardner E, Venkataraman AP, Dominguez-Vicent A, Kokkali E, Rho S, Johannesson G, Burgess RW, Fuerst PG, Brautaset R, Kolko M, Morgan JE, Crowston JG, Votruba M, Williams PA. Nicotinamide provides neuroprotection in glaucoma by protecting against mitochondrial and metabolic dysfunction. Redox Biol. 2021 Jul;43:101988. doi: 10.1016/j.redox.2021.101988. Epub 2021 Apr 24. PMID 33932867
- [Background] Verdin E. NAD(+) in aging, metabolism, and neurodegeneration. Science. 2015 Dec 4;350(6265):1208-13. doi: 10.1126/science.aac4854. PMID 26785480
- [Background] Weinreb RN, Aung T, Medeiros FA. The pathophysiology and treatment of glaucoma: a review. JAMA. 2014 May 14;311(18):1901-11. doi: 10.1001/jama.2014.3192. PMID 24825645
- [Background] Williams PA, Harder JM, Foxworth NE, Cochran KE, Philip VM, Porciatti V, Smithies O, John SW. Vitamin B3 modulates mitochondrial vulnerability and prevents glaucoma in aged mice. Science. 2017 Feb 17;355(6326):756-760. doi: 10.1126/science.aal0092. PMID 28209901
- [Background] Xie N, Zhang L, Gao W, Huang C, Huber PE, Zhou X, Li C, Shen G, Zou B. NAD+ metabolism: pathophysiologic mechanisms and therapeutic potential. Signal Transduct Target Ther. 2020 Oct 7;5(1):227. doi: 10.1038/s41392-020-00311-7. PMID 33028824
- [Background] Zapata-Perez R, Wanders RJA, van Karnebeek CDM, Houtkooper RH. NAD+ homeostasis in human health and disease. EMBO Mol Med. 2021 Jul 7;13(7):e13943. doi: 10.15252/emmm.202113943. Epub 2021 May 27. PMID 34041853
- [Background] Zhang X, Zhang N, Chrenek MA, Girardot PE, Wang J, Sellers JT, Geisert EE, Brenner C, Nickerson JM, Boatright JH, Li Y. Systemic Treatment with Nicotinamide Riboside Is Protective in Two Mouse Models of Retinal Ganglion Cell Damage. Pharmaceutics. 2021 Jun 16;13(6):893. doi: 10.3390/pharmaceutics13060893. PMID 34208613